CLINICAL TRIAL: NCT05510635
Title: The Effectiveness of Bibliotherapy on Improving Emotional Distress and Coping Strategies and Enhancing Resilience of Adolescents With Cancer: A Randomized Controlled Trial
Brief Title: The Effectiveness of Bibliotherapy on Emotional Distress, Coping Strategies and Resilience of Adolescents With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: T-24142-54260-19890
Record Dates: First submitted 2022-08-14; First posted 2022-08-22 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-08

CONDITIONS: Emotional Distress; Pediatric Cancer
Keywords: adolescent; bibliotherapy; emotional distress; coping; resilience
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interactive bibliotherapy (Experimental): All adolescents enrolled in the experimental group will receive two times of interactive bibliotherapy with an interval of 7 to 14 days. The researcher will read the story to the participant and then discuss it with him/her.
  Interventions: Other: interactive bibliotherapy
- reading bibliotherapy (Active Comparator): All adolescents enrolled in the comparison group will receive two times of reading bibliotherapy with an interval of 7 to 14 days. The participant will read the story alone.
  Interventions: Other: reading bibliotherapy

INTERVENTIONS:
Other: interactive bibliotherapy — The researcher selected two picture books whose central issues are about the common emotional distress of adolescents with cancer, that is, negative emotion coping, and self-worth. The researcher will read the story to the participant and then use the interview guideline to discuss it with him or her one by one. The interview guideline for interactive bibliotherapy is listed according to the mechanism of bibliotherapy, including identification, catharsis, and insight, and additional questions leading a reader to think deeply.
  Arms: interactive bibliotherapy
Other: reading bibliotherapy — The researcher selected two picture books whose central issues are about the common emotional distress of adolescents with cancer, that is, negative emotion coping, and self-worth. The participant can take 20 to 25 minutes to read the story. No one can bother the participant during the intervention.
  Arms: reading bibliotherapy

SUMMARY:
Adolescents with cancer who were diagnosed within two years suffered severe emotional distress. Bibliotherapy therapy uses healing materials as a medium to enable individuals experiencing emotional distress to obtain emotional healing through story situations, thereby enhancing resilience. However, there is a lack of research on bibliotherapy in adolescents with cancer. Therefore, the investigators would like to evaluate the effectiveness of interactive bibliotherapy in improving emotional distress and coping strategies and enhancing the resilience of adolescents with cancer compared to reading bibliotherapy.

DETAILED DESCRIPTION:
A multicenter randomized controlled trial will be conducted. Adolescents aged 10 to 19 years and diagnosed with cancer or relapse during the first two years will be included in the study. Seventy participants from three medical centers in northern Taiwan will be assigned to experimental or comparison groups through blocked randomization. The experimental group will receive the interactive bibliotherapy twice, and the comparison group will receive the reading bibliotherapy twice. The Positive and Negative Affect Schedule, Pediatric Cancer Coping Scale, and Haase Adolescent Resilience in Illness Scale will be used to measure participants' emotional distress, coping strategies and resilience at the time points of pre-intervention, after the intervention, and follow-up for a month after the intervention. An interview will be conducted over the intervention for a month. The generalized estimating equation will be used to analyze the two groups' emotional distress, coping strategies, and resilience. The content analysis will be performed to analyze the interview data. It is hoped that the results of this study can prove that bibliotherapy has the potential to improve emotional distress and coping strategies and enhance resilience in adolescents with cancer. This study is expected to provide health providers with novel evidence on the effectiveness of an intervention to take care of patients with cancer. Furthermore, this study provides an interdisciplinary intervention of nursing and other domain, and it may be extended to further research to improve patient care quality through cross-disciplinary coordination.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 10 to 19 years.
* Adolescents were diagnosed with leukemia or osteosarcoma.
* Adolescents were diagnosed with cancer or relapsed during the first two years.
* Adolescents who have received cancer treatment.
* Adolescents who can read picture books and communicate with Chinese.

Exclusion Criteria:

* Adolescents who have psychiatric history.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
emotional distress | Changes from Baseline to Post-Intervention and 1-month follow-up.
  The Positive and Negative Affect Schedule will be used to measure participants' emotional distress. The Positive and Negative Affect Schedule is composed of a 20-item questionnaire separated into two subscales, positive and negative affect. Each item is assessed on a 5-point Likert scale, varying from 1 to 5, obtaining total points ranging from 10 to 50 on each subscale. Higher scores suggest higher levels of positive or negative affect.
coping strategies | Changes from Baseline to Post-Intervention and 1-month follow-up.
  The Pediatric Cancer Coping Scale (PCCS) will be used to measure participants' coping strategies. The PCCS is composed of a 33-item questionnaire separated into three subscales, including cognitive coping (14 items), problem-oriented coping (9 items), and defensive coping (10 items). The PCCS is also separated into two parts. The first part of the scale is used to measure the usage frequency of each item, and the second part evaluates the efficacy of each strategy. Each item is assessed on a 4-point Likert scale, varying from 0 to 3. The score for each subscale is calculated by adding all corresponding item scores. Higher scores represent the higher usage frequency of strategies or the more effective coping strategies.
resilience | Changes from Baseline to Post-Intervention and 1-month follow-up.
  The Haase Adolescent Resilience in Illness Scale will be used to measure participants' resilience. The Haase Adolescent Resilience in Illness Scale is composed of a 13-item questionnaire. Each item is assessed on a 6-point Likert scale, varying from 1 to 6, obtaining total points ranging from 13 to 78, with higher scores representing higher resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu TJ, Sheih CS, Jou ST, Lee CY, Yu TY, Liu CY, Chen CW. Effects of bibliotherapy on emotional distress, coping strategies, and resilience in adolescents with cancer: A pilot randomized controlled trial. Eur J Oncol Nurs. 2025 Jun;76:102900. doi: 10.1016/j.ejon.2025.102900. Epub 2025 May 10. PMID 40381380